CLINICAL TRIAL: NCT01238796
Title: A Phase 1 Open-Label Study to Evaluate the Effect of Renal Function on the Biological Activity of Telavancin
Brief Title: A Study to Evaluate the Effect of Renal Function on the Biological Activity of Telavancin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9809-CL-1407
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Kidney Diseases; End Stage Renal Disease
Keywords: telavancin; Pharmacokinetics; Severe renal disease; VIBATIV®; ASP9809
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic | interventions — telavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal renal function (Experimental): Subjects with normal renal function
  Interventions: Drug: telavancin
- Severe renal impairment (Experimental): Subjects with severe renal impairment
  Interventions: Drug: telavancin
- End stage renal disease (Experimental): Subjects with end stage renal disease
  Interventions: Drug: telavancin

INTERVENTIONS:
Drug: telavancin — Intravenous
  Other Names: VIBATIV®; TD-6424; ASP9809

SUMMARY:
The purpose of this study is to evaluate the effect of renal function on the biological activity of telavancin using blood samples obtained from subjects with normal renal function, severe renal impairment, and end stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Weighs at least 45 kg and body mass index of 18 to 40 kg/m2, inclusive
* An estimated creatinine clearance value based on Cockcroft-Gault method of:

  * >80 mL/min for subjects with normal renal function
  * <30 mL/min for subjects with severe renal impairment
  * receiving hemodialysis three times a week for subjects with end stage renal impairment
* If female, the subject is at least 2 years postmenopausal, surgically sterile or practicing effective birth control, and is not pregnant or lactating
* Good venous access

Exclusion Criteria:

* History of any clinically significant acute illness (other than renal disease and conditions related to the renal disease in renal impairment subjects, such as stable diabetes or hypertension)
* Has had a kidney transplant that is still functioning
* History of unexplained syncope, cardiac arrest, unexplained cardiac arrythmia or torsade de pointes, structural heart disease, prolonged QT interval, or family history of long QT syndrome
* Known hypersensitivity to telavancin or any of the excipients in the formulation, or a history of severe allergic or anaphylactic reactions
* History of consuming more than 7 units of alcoholic beverages per week, or history of alcoholism or substance abuse within past 2 years
* Known to be positive for human immunodeficiency virus antibody
* For subjects with normal renal function, has had treatment with prescription or non-prescription drugs, including complementary and alternative medicines or over-the counter medications, with the exception of oral contraceptives, hormone replacement therapy, daily aspirin, and occasional use of acetaminophen within the past 14 days
* For subjects with renal impairment, has not been on a stable dose of concomitant medications for at least 2 weeks prior to study start or is taking any medication that would interfere with the evaluation of televancin in this study
* Has received an experimental agent within 30 days or ten half-lives, whichever is longer, prior to study drug administration
* Has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Concentration of telavancin as estimated by antibiotic potency bioassay | Days 1-4
Concentration of telavancin as determined by standard Liquid Chromatography Tandem Mass Spectrometer (LC/MS/MS) | Days 1-4

SECONDARY OUTCOMES:
Pharmacokinetic variables through analysis of blood samples | Days 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - New Orleans Center for Clinical Research, Knoxville, Tennessee